CLINICAL TRIAL: NCT01387997
Title: Nano-mechanical and Nano-electrosensing Devices Based Interaction Force and Interaction Kinetics Analysis of Oncogenic Human Papilloma Viruses
Brief Title: e- Ab Sensor-based Real-time Detection of Oncogenic Human Papilloma Viruses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 201005076R
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Cervical Cancer; Human Papilloma Virus Infection
Keywords: HPV
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: Electrosensing antibody probing system (e- Ab sensor)

INTERVENTIONS:
Device: Electrosensing antibody probing system (e- Ab sensor) — Electrosensing antibody probing system (e- Ab sensor), which was developed for the rapid and sensitive detection of hapten, proteins, or viral antigen in medical samples, will be used for analyzing the interaction kinetics between anti-high risk HPV and its antigen (high-risk HPV) present in patients. The system incorporates the use of engineered semiconducive antibodies or virus in vertical and lateral chip (eAbchip) or lateral flow through (eAbsignal) formats. In electrosensing antibody probing, semiconductive antibodies are bound as a suitable electrosensing probe, which specifically and selectively binds targeted molecules (high-risk HPV) in the test specimens. From assessment of the electric signature of semiconductive anti- high-risk HPV antibodies, the eABprobe could offer sensitive detection and precise quantification of high-risk HPV.

SUMMARY:
To develop a real-time diagnostic technique with e- Ab sensor for high risk human papilloma viruses(high risk HPV) detection, the investigators conduct a prospective clinical study. In comparison with results from direct sequencing of HPV, the investigators evaluate the performance of e- Ab sensor, including reproducibility, sensitivity, specificity, and cross-reaction (such as detection of low risk HPV). The potential factors which may interfere with the results would be investigated. With such a real-time diagnostic technique, the investigators hope to obtain information of patients in cost-saving and time-saving way and can give patients early treatment and offer more individualized treatment for our patients.

DETAILED DESCRIPTION:
Human papillomavirus (HPV)-induced cervical carcinogenesis is proposed to be multi-step in nature. The major steps in cervical carcinogenesis include persistent infection of the metaplastic cervical epithelium with one or more of the oncogenic HPV infection, clonal progression of the infected epithelium to cervical precancer, and further invasion. Although these fundamental steps are well established, several new genetic and immunologic studies have shed light on the factors that influence each of these transitions. Over 150 different HPV subtypes have been identified so far, with a subset of these being classified as high risk for oncogenesis. Persistent infection with oncogenic HPV is the main cause of cervical cancer. Polymerase-chain-reaction (PCR)-based assays show that HPV DNA exist in around 90.7- 96.6% patients with cervical cancer and in 13.4 -15.6% control women. About the detected HPV types in patients, in descending order of frequency, are types 16, 18, 45, 31, 33, 52, 58, and 35. Fifteen HPV types are classified as high-risk types (16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 68, 73, and 82); 3 are classified as probable high-risk types (26, 53, and 66); and 12 are classified as low-risk types (6, 11, 40, 42, 43, 44, 54, 61, 70, 72, 81). The most frequently detected high risk HPV types (HPV 16, 51, 52, and 59) are similar in male of different sites, which is compatible with the female incidence.

Electrosensing antibody probing system (e- Ab sensor), which was developed for the rapid and sensitive detection of hapten, proteins, or viral antigen in medical samples, will be used for analyzing the interaction kinetics between anti-high risk HPV and its antigen (high-risk HPV) present in patients. The system incorporates the use of engineered semiconducive antibodies or virus in vertical and lateral chip (eAbchip) or lateral flow through (eAbsignal) formats. In electrosensing antibody probing, semiconductive antibodies are bound as a suitable electrosensing probe, which specifically and selectively binds targeted molecules (high-risk HPV) in the test specimens. From assessment of the electric signature of semiconductive anti- high-risk HPV antibodies, the eABprobe could offer sensitive detection and precise quantification of high-risk HPV.

To develop a real-time diagnostic technique with e- Ab sensor for high risk HPV detection, the investigators conduct a prospective clinical study. In comparison with results from direct sequencing of HPV, the investigators evaluate the performance of e- Ab sensor, including reproducibility, sensitivity, specificity, and cross-reaction (such as detection of low risk HPV). The potential factors which may interfere with the results would be investigated. e- Ab sensor threshold decisions must maximize its sensitivity. Therefore, the threshold value in the test group is to find the decision could have 90% sensitivity and 90% specificity.With such a real-time diagnostic technique, the investigators hope to obtain information of patients in cost-saving and time-saving way and can give patients early treatment and offer more individualized treatment for our patients.

ELIGIBILITY:
Inclusion Criteria:

* A:The patients with confirmed or suspected infection.
* B: The patients without disease.

Exclusion Criteria:

* The patients with chronic diseases or medical disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2010-06; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The performance of e- Ab sensor | 1 Day
  In comparison with results from direct sequencing of HPV, we evaluate the performance of e- Ab sensor, including reproducibility, sensitivity, specificity, and cross-reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Bor-Ching Sheu, MD,PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan